CLINICAL TRIAL: NCT01891656
Title: In-Person VS. Computer Interventions for Increasing Probation Compliance
Brief Title: Motivational Assessment Program to Initiate Treatment
Acronym: MAPIT
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of North Texas Health Science Center (Other)
Collaborators: National Institute on Drug Abuse (NIDA) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: R01DA029010-01 (NIH); 5R01DA029010-06 (NIH)
Record Dates: First submitted 2011-10-18; First posted 2013-07-03 (Estimated); Last update posted 2016-04-13 (Estimated); Status verified 2016-04

CONDITIONS: Substance-Related Disorders
Keywords: Motivational Interviewing; Internet; Treatment; Substance-Related Disorders; Criminal Justice
MeSH Terms: conditions — Substance-Related Disorders | interventions — Motivational Interviewing

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (3):
- Motivational Interviewing (Experimental): Participants randomized to the MI group will receive a single 60-minute MI session focused on motivation to initiate and engage in treatment. The MI session will be organized around the "Check-Up" format, with additional planning components as desired by the client.
  Interventions: Behavioral: Motivational Interviewing
- Supervision As Usual (No Intervention): Participants randomized to the SAU group will receive the standard agency intake process as well as baseline and follow-up research interviews, but will not receive any additional intervention as part of the study. They will be referred to a treatment program as per the normal routine.
- Motivational Computer (Experimental): Participants randomized to the MC group will complete a 60 minute computer intervention focused on motivation to initiate and engage in treatment. The program will be self-guided, interactive, and to the extent possible, will mirror the features of MI session. The MC program will have two main components: a motivation component and a planning component.
  Interventions: Behavioral: Motivational Computer

INTERVENTIONS:
Behavioral: Motivational Interviewing — MI is a "client centered, directive style of interacting with a person to help explore and resolve ambivalence about change" (Miller & Rollnick, 2002). MI borrows from Client-Centered Counseling in its emphasis on empathy, optimism, and respect for client choice (Rogers, 1961). MI also draws from Self-Perception Theory, which says that a person becomes more or less committed to an action based on the verbal stance he or she takes (Bem, 1972). The effects of MI tend to be in the small-to-medium range when compared to no treatment, and nonsignificant when compared to more extensive treatment.
  Other Names: Motivational Enhancement Therapy
  Arms: Motivational Interviewing
Behavioral: Motivational Computer — The growing use of technology has led to the development of automated interventions for behavior change, including some that target drug and alcohol use (Elliott, et al, 2008; Lustria, et al, 2009; Revere & Dunbar, 2001; Walters, et al, 2006) and treatment interest (Lieberman & Massey, 2008). As discussed by Hester & Miller (2006), automated interventions have several potential advantages over face-to-face interventions: (I) They require little or no staff contact, which may increase cost-effectiveness; (2) they can allow for automatic data collection and follow-up; and (3) they can be disseminated with little loss of fidelity.
  Other Names: Web-Based Interventions
  Arms: Motivational Computer

SUMMARY:
Substance abuse treatment in the criminal justice system can reduce drug use and related criminal behavior. Although drug and alcohol treatment are common mandates in criminal justice programs, only a minority of clients actually initiate treatment. This proposal will compare two intervention formats that target motivation to initiate and engage in treatment among a group of probationers who have drug or alcohol treatment conditions. Six hundred drug and alcohol offenders in two probation sites (Baltimore, MD and Dallas, TX) will be randomized to receive: 1) an in-person motivational interviewing session (MI), 2) a motivational computer program (MC), or 3) supervision intake and monitoring as usual (SAU). The MI condition will be structured along the lines of the "Check-Up" format which consists of an assessment and personalized feedback delivered in an MI style; the content of the MC condition will be drawn from previous literature on effective motivational computer programs. Both interventions will be delivered at the start of the probation process, with follow-up assessments at 2 and 6 months. Primary outcomes include engagement and participation in substance abuse treatment; secondary outcomes include drug and alcohol use, probation progress, criminal behavior, and HIV testing and care. This project will be the first to develop and test two interventions for encouraging criminal justice clients to follow through with treatment recommendations, with the goal of increasing treatment initiation, and reducing subsequent drug use and criminal behavior. It also contributes to ongoing partnerships with two large probation agencies-the Dallas County Supervision and Corrections Department and the Maryland Division of Parole and Probation.

DETAILED DESCRIPTION:
Specific Aims

* Develop two intervention formats (Motivational Interviewing (MI) and Motivational Computer (MC)) for increasing motivation to initiate and engage in substance abuse treatment and/or HIV / AIDS testing and, if appropriate, HIV care.
* Test the efficacy of MI and MC on treatment initiation and participation, substance abuse, HIV testing/care, and recidivism, as compared to Supervision As Usual (SAU);
* Evaluate offender characteristics (e.g., risk level, gender, ethnicity, motivation) as potential moderators of the intervention effect; and,
* Assess the relative cost and cost-effectiveness of MI and MC on substance abuse treatment and/or linkage to or participation in HIV/AIDS care, supervision outcomes, recidivism, and substance abuse.

ELIGIBILITY:
Inclusion Criteria:

* >=18 years old
* Drug or Alcohol use in the last 90 days

Exclusion Criteria:

* <18 years old
* Cannot speak English
* Already participate in a substance abuse treatment

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 380 (Actual)
Dates: Start 2012-06; Primary Completion 2015-06 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
Treatment Progress | 6 months
  Treatment progress assesses initiation, engagement and retention at 2 and 6 months via telephone. In-person visits are assessed at baseline and during a 6 month visit.

SECONDARY OUTCOMES:
Drug and Alcohol Use | 6 months
  Drug and alcohol use is a secondary outcome measured at baseline and 6 months during an in-person interview. In addition, this outcome is measured at 2 via telephone.
Probation Progress | 6 months
  Probation progress is measured at baseline and 6 months via in-person interview. In addition, this outcome is measured at 2 via a telephone interview.
Criminal Behavior | 6 months
  Criminal Behavior is measured during in-person interviews at baseline and 6 months. In addition, this outcome is measured at 2 months via telephone.

CONTACTS AND LOCATIONS:
Overall Officials: Scott T Walters, PhD, Principal Investigator — UNT Health Science Center
Locations (2):
- United States (2):
  - University of North Texas Health Science Center, Fort Worth, Texas
  - George Mason University, Fairfax, Virginia

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Walters ST, Ondersma SJ, Ingersoll KS, Rodriguez M, Lerch J, Rossheim ME, Taxman FS. MAPIT: development of a web-based intervention targeting substance abuse treatment in the criminal justice system. J Subst Abuse Treat. 2014 Jan;46(1):60-5. doi: 10.1016/j.jsat.2013.07.003. Epub 2013 Aug 16. PMID 23954392
- [Result] Reingle Gonzalez JM, Walters ST, Lerch J, Taxman FS. The Relationship Between Drug Use, Drug-related Arrests, and Chronic Pain Among Adults on Probation. J Subst Abuse Treat. 2015 Jun;53:33-8. doi: 10.1016/j.jsat.2014.12.005. Epub 2014 Dec 30. PMID 25595302
- [Derived] Rodriguez M, Walters ST, Houck JM, Ortiz JA, Taxman FS. The language of change among criminal justice clients: Counselor language, client language, and client substance use outcomes. J Clin Psychol. 2018 Apr;74(4):626-636. doi: 10.1002/jclp.22534. Epub 2017 Sep 22. PMID 28940435
- [Derived] Lerch J, Walters ST, Tang L, Taxman FS. Effectiveness of a computerized motivational intervention on treatment initiation and substance use: Results from a randomized trial. J Subst Abuse Treat. 2017 Sep;80:59-66. doi: 10.1016/j.jsat.2017.07.002. Epub 2017 Jul 6. PMID 28755774
- [Derived] Spohr SA, Taxman FS, Rodriguez M, Walters ST. Motivational Interviewing Fidelity in a Community Corrections Setting: Treatment Initiation and Subsequent Drug Use. J Subst Abuse Treat. 2016 Jun;65:20-5. doi: 10.1016/j.jsat.2015.07.012. Epub 2015 Jul 29. PMID 26365536
- [Derived] Taxman FS, Walters ST, Sloas LB, Lerch J, Rodriguez M. Motivational tools to improve probationer treatment outcomes. Contemp Clin Trials. 2015 Jul;43:120-8. doi: 10.1016/j.cct.2015.05.016. Epub 2015 May 22. PMID 26009023